CLINICAL TRIAL: NCT00003635
Title: A Multicenter Study to Assess the Efficacy of 506U78 in Patients With Chronic Lymphocytic Leukemia Who Are Refractory to Fludarabine and Alkylator Therapy
Brief Title: 506U78 in Treating Patients With Chronic Lymphocytic Leukemia That Has Not Responded to Fludarabine or Alkylating Agents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: GW-PGAA2003; CDR0000066719 (Registry Identifier: PDQ (Physician Data Query)); CWRU-GLAX-1999; MB-405; NCI-98-C-0164; UCLA-991004701A
Record Dates: First submitted 1999-11-01; First posted 2004-03-31 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2002-01

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic | interventions — nelarabine

INTERVENTIONS:
Drug: nelarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of 506U78 in treating patients with chronic lymphocytic leukemia that has not responded to fludarabine or alkylating agents.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the anticancer efficacy of 506U78 in patients with chronic lymphocytic leukemia refractory to fludarabine and alkylator therapy. II. Determine the safety (including incidence of infection) of this drug in these patients. III. Evaluate the pharmacokinetics of 506U78 and ara-G, and assess the intracellular pharmacokinetics of ara-GTP in patients receiving multiple treatment courses (at M.D. Anderson Cancer Center only). IV. Determine the response rate, time to maximal response, and duration of response in patients treated with this drug. V. Determine two-year survival and progression-free survival of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to cellular type of disease (B cell vs T cell). Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Treatment repeats every 28 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at 28 days and then every 2 months for 2 years until disease progression. After disease progression, patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: Approximately 14-100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of refractory chronic lymphocytic leukemia Evidence of active disease after fludarabine or alkylator therapy Must meet one or more of the following criteria for active disease: Minimum of one of the following disease-related symptoms: Weight loss of 10% or more within the previous 6 months Extreme fatigue (e.g., unable to work or perform usual activities) Fevers greater than 100.5 degrees F for 2 weeks or more without evidence of infection Night sweats without evidence of infection Evidence of progressive marrow failure manifested by the development or worsening of autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroid therapy Massive (e.g., greater than 6 cm below the left costal margin) or progressive splenomegaly Massive nodes or clusters (e.g., greater than 10 cm in longest diameter) or progressive lymphadenopathy Progressive lymphocytosis with an increase of more than 50% over a 2-month period or an anticipated doubling time of less than 6 months Ineligible if marked hypogammaglobulinemia or development of monoclonal protein in the absence of the above criteria for active disease Must have one of the following resulting from prior fludarabine or alkylator-containing therapy: Disease progression during therapy Failure to respond or obtained less than a partial response to therapy Disease progression within 6 months of the last course of therapy after an initial response Failure to respond or disease progression allowed at any time after the final dose if alkylator agent was not the most recent therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 12 weeks Hematopoietic: See Disease Characteristics Hepatic: See Disease Characteristics Bilirubin no greater than 2 times upper limit of normal No liver dysfunction due to organ infiltration by lymphocytes Renal: Creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for up to 28 days after study No neurotoxicity of grade 2 or higher No history of significant neurologic toxicity (grade 2 or greater motor or sensory impairment) due to prior chemotherapy or radiotherapy No history of seizure disorder No active infection No other malignancy within the past 2 years (except adequately treated non- melanomatous skin cancer or carcinoma in situ) that would preclude study No systemic nonmalignant comorbid disease that would preclude study No psychological, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow or peripheral blood stem cell transplantation Recovered from prior immunotherapy At least 4 weeks since prior biologic therapy and recovered Concurrent growth factors allowed Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered No prior 506U78 therapy No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics No concurrent corticosteroid therapy greater than 10 mg/day of prednisone equivalent No concurrent corticosteroids as antiemetics Concurrent hormone replacement therapy or oral contraceptives allowed Concurrent hydrocortisone as prophylaxis or treatment of transfusion reactions allowed Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonya M. Peele, MS, Study Chair — GlaxoSmithKline
Locations (22):
- United States (22):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Scripps Clinic, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - Clinical Studies, Ltd., Denver, Colorado
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Greenville Hospital System, Greenville, South Carolina
  - Physician Reliance Network, Inc., Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas